CLINICAL TRIAL: NCT02325206
Title: Randomized, Double-blind, Placebo-controlled, Single-center Phase 1 Study to Explore the Safety and Pharmacokinetics of DAPAglifozin as Add-on to Intravenous Insulin-infusion in Adolescents and Adults With Type 1 Diabetes
Brief Title: Phase 1 Study to Explore the Safety and Pharmacokinetics of DAPAglifozin in Adolescents and Adults With Type 1 Diabetes
Acronym: DAPA-IIT1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Principal Investigator, Thomas Danne, Prof. Dr. med., Kinderkrankenhaus auf der Bult
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-14-10179
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dapafliflozin (Experimental): one administration of 10mg dapagliflozin as tablet
  Interventions: Drug: dapagliflozin
- placebo (Placebo Comparator): one administration as tablet identical to the experimental drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dapagliflozin — one administration in the morning
  Other Names: Forxiga
  Arms: dapafliflozin
Drug: Placebo — one administration in the morning
  Other Names: Control
  Arms: placebo

SUMMARY:
Dapagliflozin has been effective at lowering glucose and hemoglobin A1c (HbA1C) in subjects with tpye 2 diabetes (T2DM), when studied as monotherapy as well as in combination with insulin or oral anti-diabetic medications.This lead to investigations if this therapy would also be of benefit in type 1 diabetes as intensive insulin therapy is associated with glucose fluctuations, hypoglycemia, weight gain, and subsequent insulin resistance, all of which may reduce efficacy.

The purpose of the pilot study is to collect clinical data on the HbA1c-dependent effect of a single-dose of 10mg dapagliflozin on the insulin dose administered intravenously during a glucose-infusion and an oral mixed-meal for the ensuing 24 hours with blood glucose kept between 160 - 220 mg/dl.

The first objective is to investigate the degree of insulin dose reduction 24 hours after a single dose of 10mg dapagliflozin in patients with type 1 diabetes Further objectives are to investigate

* the effect on urinary glucose excretion
* if this effect is influenced by baseline glycemic control
* if dapagliflozin influences postprandial insulin need
* if dapagliflozin is associated with elevated ß-hydroxybutyrate levels
* PK after oral administration of 10mg dapagliflozin

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety profile and tolerability, particularly with regard to hypoglycemia and ketone development, following once daily oral dose of 10 mg of dapagliflozin administered in subjects with type 1 diabetes (T1DM) as a single dose as well as pharmacokinetics (PK) for 18 hours of treatment.

The study aimed to patients who have different degrees of inadequate glycemic control despite insulin use. Approximately 36 subjects will be screened in order to randomize 10 patients in each different HbA1C category.

The trial will consist of six visits: a screening visit (Visit 1), two dosing visits (Visit 2 and Visit 4), two phone visits (Visit 3 and Visit 5) and a follow-up visit (Visit 6). Furthermore, an information visit will take place prior to the screening visit in order to obtain patient's informed consent. Screening will take place 2-21 days prior to Visit 2 and the follow-up visit will take place 5-21 days after the end of Visit 4. The dosing visits will be separated by a wash-out period (5-30 days between the end of Visit 2 and begin of Visit 4) during which the subjects will resume their normal insulin treatment. Each phone visit (Visit 3 and Visit 5) will take place 3-5 days after the end of dosing Visits 2 and 4. The planned total duration of the trial is 18-78 days per subject (rescheduled visits excluded). Each subject will be randomised to a treatment sequence consisting of two treatment periods in which the subjects will receive dapagliflozin and placebo on two separate dosing visits.

Subjects metabolic control will be achieved by a variable i.v. infusion of human insulin by an infusion pump. The procedure will be used in order to aim and maintain blood glucose levels between 160 and 220 mg/dl thereby being in the range of the urinary threshold of glucose.

The fluid infusion and insulin dosing scheme will depend on body weight (BW) and blood glucose (BG) levels.

Two standardized mixed-meals will be given 6 hours and 12 hours after dosing. Blood glucose measurements will be performed every 15min for 120min after the mixed-meal.

Blood samples for determination of dapagliflozin concentration in serum will be taken 18times in 24hours as well as every urine sample will be collected for 24 hours after dosing for the determination of 24hour urinary glucose and creatinine for efficacy measurement.

After conclusion of the trial the documented insulin doses over time will be summed up for calculation of the total insulin dose and the insulin dose per kg body weight per 24 hours. Separate calculations will be done for the overnight period pre-dosing, six hours after dosing, two hours prior and after the first and second Standard Meal and until the end of the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent from participant and all legal representatives prior to any study specific procedures
2. Female and/or male aged 12 to 21years (both inclusive)
3. Subject must have type 1 diabetes (as diagnosed clinically) ≥ 12months
4. without completely inadequate glycemic control, defined as local laboratory A1c above 12.5% (subjects will be stratified according to glycemic control being in target (A1c 5.5 to 7.4%), slightly elevated (7.5 - 9.0%) or clearly elevated 9.1 - 12.5% ) obtained at the screening visit (Note: A one-time central laboratory re-test of the A1C is allowed)
5. Insulin use with an average daily dose between 0.6 - 2.0 U/kg, either continuous subcutaneous insulin infusion, (CSII) or multiple doses (at least 2x/day) of insulin
6. BMI 18.0 to 35.0 kg/m2 for adults or BMI between 10th and 99th age and gender related centile for pediatric patients
7. Minimum weight of 50 kg
8. Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy throughout the study as judged by the investigator
9. WOCBP must have a negative urine pregnancy test at screening as well as at Visit 2 and Visit 4.
10. Women must not be breastfeeding

Exclusion Criteria:

1. History of T2DM, maturity onset diabetes of young (MODY), pancreatic surgery or chronic pancreatitis
2. Any use of oral hypoglycemic agents within 12 months prior to the screening visit
3. History of diabetes ketoacidosis (DKA) within 12 weeks prior to prior to the screening visit
4. History of diabetes insipidus
5. History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 3 months prior to prior to the screening visit
6. Frequent episodes of hypoglycemia as defined by more than one episode requiring assistance, emergency care (paramedics or emergency room care) or glucagon therapy, or more than 2 unexplained episodes of symptomatic hypoglycemia within 3 months prior to the screening visit. An unexplained event is defined as an event that cannot be explained by circumstances such as dietary (e.g. missed meal), strenuous exercise, error in insulin dosing, etc.
7. Hypoglycemic unawareness
8. History of Addison's disease or chronic adrenal insufficiency
9. Prisoners or subjects who are involuntarily incarcerated
10. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
11. Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid taken for > 4 weeks within 3 months prior to Day -3 visit. NOTE: Topical or inhaled corticosteroids are allowed.
12. Any unstable endocrine, psychiatric, rheumatic disorders as judged by the Investigator.
13. Subject is, in the judgment of the Investigator, unlikely to comply with the protocol or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data.
14. Subject with any condition which, in the judgment of the Investigator, may render the subject unable to complete the study or which may pose a significant risk to the subject.
15. Subject is currently abusing alcohol or other drugs or has done so within the last 6 months.
16. Subject is a participating investigator, study coordinator, employee of an investigator or immediate family member of any of the aforementioned.
17. Administration of any other investigational drug within 30 days of planned enrolment to this study.
18. No clinical conditions or clinically significant abnormalities, in any laboratory value(s) collected after screening and prior to randomization which, in the Investigator's judgment, should preclude entry into the treatment period

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
reduction of intravenous insulin dose | 24hours
  reduction of intravenous insulin dose with glucose kept between 160 - 240 mg/dl 24 hours after oral administration of 10mg dapagliflozin

SECONDARY OUTCOMES:
HbA1c effect | 24hours
  effect of baseline HbA1c on insulin-dose lowering effect of 10mg dapagliflozin
urinary glucose excretion | 24hours
  increase of urinary glucose excretion with blood glucose kept between 160 - 220 mg/dl 24 hours after oral administration of 10mg dapagliflozin

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Danne, MD, Principal Investigator — Kinderkrankenhaus auf der Butl
Locations (1):
- Kinder - und Jugendkrankenhaus AUF DER BULT, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No